CLINICAL TRIAL: NCT02421601
Title: A Multicenter, Open-label Study of SI 6603 in Patients With Lumbar Disc Herniation (Phase III)
Brief Title: A Study of SI-6603 in Patients With Lumbar Disc Herniation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seikagaku Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6603/1132
Record Dates: First submitted 2015-04-06; First posted 2015-04-20 (Estimated); Results first posted 2021-11-11 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Intervertebral Disc Disease; Lumbar Disc Disease
MeSH Terms: conditions — Intervertebral disc disease

ARMS (1):
- SI-6603 (Experimental): SI-6603: SI-6603 is administrated into the nucleus pulposus of the intervertebral disc
  Interventions: Drug: Condoliase

INTERVENTIONS:
Drug: Condoliase — 1.25 U, intradiscal injection, one time

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of SI-6603(Condoliase) in patients with lumbar disc herniation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lumbar disc herniation (L1-L2, L2-L3, L3-L4, L4-L5 or L5-S1) as assessed by MRI and clinical symptoms corresponding to position of the impaired nerve root.
* Patients assessed as positive in the Femoral Nerve Stretching (FNS) test for L1-L2, L2-L3, or L3-L4 and Straight Leg Raising (SLR) test.
* Patients with sciatica in either leg.
* Patients with no improvement from conservative treatment

Exclusion Criteria:

* Patients who have 2 or more lumbar disc herniations as assessed by MRI.
* Patients in whom a rupture into the posterior longitudinal ligament is identified by MRI.
* Patients who have undergone lumbar operation, or lumbar percutaneous nucleotomy or lumbar intradiscal therapies

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1011 (Actual)
Dates: Start 2015-03; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (30):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Gold River, California
  - Laguna Hills, California
  - Los Gatos, California
  - Riverside, California
  - Temecula, California
  - Greenwood Village, Colorado
  - Clermont, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Miami Gardens, Florida
  - Naples, Florida
  - Pinellas Park, Florida
  - Sarasota, Florida
  - South Miami, Florida
  - St. Petersburg, Florida
  - Winter Park, Florida
  - Marietta, Georgia
  - Newnan, Georgia
  - Bloomington, Illinois
  - Carmel, Indiana
  - Shreveport, Louisiana
  - City of Saint Peters, Missouri
  - Hartsdale, New York
  - Eugene, Oregon
  - Charleston, South Carolina
  - Plano, Texas
  - Sandy City, Utah
- Germany (6):
  - Eichstätt, Bavaria
  - Frankfurt am Main, Hesse
  - Cologne, North Rhine-Westphalia
  - Göppingen, Stuttgart
  - Berlin
  - Hamburg
- Romania (3):
  - Brasov
  - Bucharest
  - Sibiu
- Spain (9):
  - Cadiz, Andalusia
  - Palma de Mallorca, Balearic Islands
  - Badalona, Barcelona
  - Terrassa, Barcelona
  - Valladolid, Castille and León
  - Alcorcón, Madrid
  - Barcelona
  - Ourense
  - Valencia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients are enrolled in the study once eligibility is determined, but after enrollment, injection to the intervertebral disc may not be feasible due to anatomical reasons and patient condition during injection procedure. Therefore, Enrollment number in the Protocol Section (1011) and patients who Started the study (991) are not necessarily the same.
Groups:
- SI-6603: Patients received a single-dose injection of SI-6603 1.25 U into an intervertebral disc.
Period: Overall Study
Arm/Group | SI-6603
Started | 991
Completed | 909
Not Completed | 82
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 5
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 31
Not completed — Others | 41

BASELINE CHARACTERISTICS:
Arm/Group | SI-6603
Number analyzed (Participants) | 991
Age, Customized [Mean (Standard Deviation); unit: years] | 49.1 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 539
  Male | 452
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 4
  Race: White | 862
  Race: Black | 103
  Race: Other | 22
Region of Enrollment [Number; unit: participants]
  United States | 824
  Germany | 70
  Spain | 75
  Romania | 22
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Number analyzed differs from overall population, due to data availability for analysis.
  kg/m^2
    number analyzed (Participants) | 989
    (all) | 29.44 (6.172)
Leg Pain (VAS) [Mean (Standard Deviation); unit: mm] — Worst leg pain intensity during the past 24 hours assessed by Visual Analog Scale (VAS). Scores are recorded by making a handwritten mark on a 100 mm line that represents a continuum between "no pain" (0 mm) and "extreme pain" (100 mm). Population: Number analyzed differs from overall population, due to data availability for analysis.
  mm
    number analyzed (Participants) | 990
    (all) | 67.9 (18.48)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAE)
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event (AE) that began or that worsened in severity after the investigational drug had been administered. All AEs, including intercurrent illnesses and regardless of the relationship to investigational drug, occurring during the study were documented from the signing of the informed consent form until completion of final visit. Concomitant illnesses, which existed before entry into the study, were not considered AEs unless they worsened during the treatment period. All AEs, regardless of the source of identification (e.g., physical examination, laboratory assessment, or reported by patient), had to be documented.
Time Frame: 26 weeks
Population: Number of Patients with at Least 1 Treatment-Emergent Adverse Event N (%)
Measure: Count of Participants; unit: Participants
Arm/Group | SI-6603
Number analyzed (Participants) | 991
Participants | 615

2. Secondary Outcome: Worst Leg Pain as Assessed by Visual Analog Scale (VAS)
Description: Worst leg pain intensity during the past 24 hours assessed by Visual Analog Scale (VAS). Scores are recorded by making a handwritten mark on a 100 mm line that represents a continuum between "no pain" (0 mm) and "extreme pain" (100 mm).
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SI-6603
Number analyzed (Participants) | 900
units on a scale | 28.6 (29.61)

ADVERSE EVENTS:
Time Frame: 26 Weeks
Arm/Group | SI-6603
All-Cause Mortality (participants affected / at risk) | 4/991
Serious Adverse Events (participants affected / at risk) | 36/991
Other Adverse Events (participants affected / at risk) | 615/991
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SI-6603 (N=991)
Pneumonia (Infections and infestations) | 1
Urinary tract infection bacterial (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hodgkin's disease recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Drug dependence (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 2
Cerebral ischaemia (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Paraspinal abscess (Musculoskeletal and connective tissue disorders) | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 1
Nuclear magnetic resonance imaging abnormal (Investigations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2
Road traffic accident (Injury, poisoning and procedural complications) | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SI-6603 (N=991)
Nuclear magnetic resonance imaging spinal abnormal (Investigations) | 206
Back pain (Musculoskeletal and connective tissue disorders) | 158
Spinal X-ray abnormal (Investigations) | 76
Pain in extremity (Musculoskeletal and connective tissue disorders) | 54
C-reactive protein increased (Investigations) | 40
Sciatica (Nervous system disorders) | 27
Arthralgia (Musculoskeletal and connective tissue disorders) | 25
Nasopharyngitis (Infections and infestations) | 20
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17
Nausea (Gastrointestinal disorders) | 15
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 14
Headache (Nervous system disorders) | 14
Sinusitis (Infections and infestations) | 13
White blood cell count increased (Investigations) | 12
Rash (Skin and subcutaneous tissue disorders) | 11
Blood triglycerides increased (Investigations) | 10
Upper respiratory tract infection (Infections and infestations) | 10
Influenza (Infections and infestations) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT02421601/Prot_SAP_000.pdf